CLINICAL TRIAL: NCT02658929
Title: CRB-401 A Phase 1 Study of bb2121 in BCMA-Expressing Multiple Myeloma
Brief Title: Study of bb2121 in Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Genetix Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRB-401
Record Dates: First submitted 2016-01-15; First posted 2016-01-20 (Estimated); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Efficacy and Safety; bb2121; CAR T Cell; BCMA
MeSH Terms: conditions — Multiple Myeloma | interventions — idecabtagene vicleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- bb2121 (Experimental): bb2121 autologous CAR T cells will be infused at a dose ranging from 150 - 450 x 10^6 CAR+ T cells after receiving lymphodepleting chemotherapy
  Interventions: Biological: bb2121

INTERVENTIONS:
Biological: bb2121 — bb2121

SUMMARY:
Study CRB-401 is a 2-part, non-randomized, open label, multi-site Phase 1 study of bb2121 in adults with relapsed/refractory multiple myeloma (MM).

DETAILED DESCRIPTION:
This is a 2-part, non-randomized, open label, multi-site Phase 1 study. the study design consists of 2 parts: Part A (Dose Escalation), in which the RP2D is determined, and Part B (Expansion Cohorts), in which subjects are treated with the determined RP2D.

Following consent, enrolled subjects will undergo a leukapheresis procedure to collect autologous mononuclear cells for manufacture of investigational drug product (bb2121). Following manufacture of the drug product, subjects will receive lymphodepleting therapy with fludarabine and cyclophosphamide prior to bb2121 infusion. All subjects who have received bb2121 infusion will be followed for up to 60 months on CRB-401.

All subjects who complete the study, as well as those who withdraw from the study after receiving bb2121 for reasons other than death or meeting the early termination criteria, will be asked to continue to undergo long-term follow-up in a companion study for up to 15 years after their last bb2121 infusion, with a focus on long-term safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age at the time of signing informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Subjects must have measurable disease including at least one of the criteria below:

Serum M-protein greater or equal to 0.5 g/dL Urine M-protein greater or equal to 200 mg/24 h Serum free light chain (FLC) assay: involved FLC level greater or equal to 10 mg/dL (100 mg/L) provided serum FLC ratio is abnormal -Women of child-bearing potential (WCBP) must have a negative serum pregnancy test prior to treatment and refrain from tissue donation including egg donation or any other tissue/blood/organ donations, for at least 1 year following bb2121 infusion. All sexually active WCBP and all sexually active male subjects must agree to use effective methods of birth control throughout the study. All sexually active males subjects must refrain from tissue donation including egg donation or any other tissue/blood/organ donations, for at least 1 year following bb2121 infusion.

Part A:

Diagnosis of MM with relapsed or refractory disease and have had at least 3 different prior lines of therapy including proteasome inhibitor (e.g., bortezomib or carfilzomib) and immunomodulatory therapy (IMiD; e.g., lenalidomide or pomalidomide), or have "double refractory" disease to a proteasome inhibitor and IMiD, defined as progression on or within 60 days of treatment with these agents

- Part B: Diagnosis of MM with relapsed or refractory disease with previous exposure to PI (e.g., bortezomib or carfilzomib), IMiDs (e.g., lenalidomide or pomalidomide), and daratumumab, and refractory (based on IMWG criteria) to their last line of therapy

Exclusion Criteria:

* Subjects with known central nervous system disease
* Inadequate hepatic function
* Inadequate renal function
* Inadequate bone marrow function
* Presence of active infection within 72 hours
* Significant co-morbid condition or disease which in the judgment of the Investigator would place the subject at undue risk or interfere with the study; examples include, but are not limited to, cirrhotic liver disease, sepsis, recent significant traumatic injury, and other conditions
* Subjects with second malignancies in addition to myeloma if the second malignancy has required therapy in the last 3 years or is not in complete remission
* Subjects with a history of class III or IV congestive heart failure or non-ischemic cardiomyopathy, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the previous 6 months
* Known human immunodeficiency virus (HIV) positivity
* Subjects who have plasma cell leukemia or clinically significant amyloidosis
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2019-07-22 (Actual); Study Completion 2022-09-22 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and abnormal laboratory test results, including dose limiting toxicities (DLTs) | Day 1 through Month 60

SECONDARY OUTCOMES:
Disease-specific response criteria including: overall response rate (ORR), complete response (CR), very good partial response (VGPR), and partial response (PR) according to the International Myeloma Working Group (IMWG) Uniform Response Criteria for MM. | Day 1 through Month 60
  Percentage of subjects who achieved a CR, VGR, PR according to IMWG Uniform Response Criteria for Multiple Myeloma (MM).

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Hege, MD, Study Director — Celgene Corporation
Locations (9):
- United States (9):
  - Stanford Cancer Center, Stanford, California
  - National Cancer Institute, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mt. Sinai Medical Center Division of Hematology/Oncology, New York, New York
  - Sarah Cannon Research Inst, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Raje N, Berdeja J, Lin Y, Siegel D, Jagannath S, Madduri D, Liedtke M, Rosenblatt J, Maus MV, Turka A, Lam LP, Morgan RA, Friedman K, Massaro M, Wang J, Russotti G, Yang Z, Campbell T, Hege K, Petrocca F, Quigley MT, Munshi N, Kochenderfer JN. Anti-BCMA CAR T-Cell Therapy bb2121 in Relapsed or Refractory Multiple Myeloma. N Engl J Med. 2019 May 2;380(18):1726-1737. doi: 10.1056/NEJMoa1817226. PMID 31042825
- [Derived] Lin Y, Raje NS, Berdeja JG, Siegel DS, Jagannath S, Madduri D, Liedtke M, Rosenblatt J, Maus MV, Massaro M, Petrocca F, Yeri A, Finney O, Caia A, Yang Z, Martin N, Campbell TB, Rytlewski J, Fuller J, Hege K, Munshi NC, Kochenderfer JN. Idecabtagene vicleucel for relapsed and refractory multiple myeloma: post hoc 18-month follow-up of a phase 1 trial. Nat Med. 2023 Sep;29(9):2286-2294. doi: 10.1038/s41591-023-02496-0. Epub 2023 Aug 17. PMID 37592106
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome